CLINICAL TRIAL: NCT02620696
Title: Effect of Netazepide, a Gastrin/CCK2 Receptor Antagonist, on Esomeprazole-induced Increases in Circulating Gastrin and Chromogranin A, and on Esomeprazole Withdrawal in Healthy Subjects
Brief Title: Effect of Netazepide on Omeprazole-induced Changes in Chromogranin A and Gastrin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-013
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: ECL-cell Hyperplasia; Parietal-cell Hyperplasia; Rebound Hyperacidity; Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — YF 476

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment 1 (Experimental): * esomeprazole 40 mg daily for 28 days (Days 1-28)
  * netazepide placebo daily from Days 1-42
  Interventions: Drug: netazepide
- Treatment 2 (Experimental): * esomeprazole 40 mg daily for 28 days (Days 1-28)
  * netazepide 25 mg daily for 14 days (Days 15-28)
  * netazepide placebo daily from Days 1-14, and from Days 29-42
  Interventions: Drug: netazepide
- Treatment 3 (Experimental): * esomeprazole 40 mg daily for 28 days (Days 1-28)
  * netazepide 25 mg daily for 14 days (Days 29-42)
  * netazepide placebo daily from Days 1-28
  Interventions: Drug: netazepide
- Treatment 4 (Experimental): * esomeprazole 40 mg daily for 28 days (Days 1-28)
  * netazepide placebo daily from Days 1-28
  Interventions: Drug: netazepide
- Treatment 5 (Experimental): * esomeprazole 40 mg daily for 28 days (Days 1-28)
  * netazepide 1 mg daily for 14 days (Days 15-28)
  * netazepide placebo daily from Days 1-14
  Interventions: Drug: netazepide
- Treatment 6 (Experimental): * esomeprazole 40 mg daily for 28 days (Days 1-28)
  * netazepide 5 mg daily for 14 days (Days 15-28)
  * netazepide placebo daily from Days 1-14
  Interventions: Drug: netazepide

INTERVENTIONS:
Drug: netazepide
  Other Names: YF476

SUMMARY:
Hypergastrinaemia induced by proton pump inhibitor (PPI) treatment is reported to cause ECL-cell and parietal-cell hyperplasia, and rebound hyperacidity and dyspepsia after PPI withdrawal.

The objective of the study was to determine the dosage regimen of netazepide, a gastrin/CCK2 receptor antagonist, required to inhibit the trophic effects of PPI-induced hypergastrinaemia.

Six groups of 8 healthy subjects participated in a randomised, double-blind, placebo-controlled exploratory study of esomeprazole 40 mg daily for 28 days, and netazepide 1, 5 or 25 mg, or placebo daily during the last 14 days of esomeprazole dosing, or 14 days after esomeprazole withdrawal. Serum gastrin and plasma chromogranin A (CgA) were measured regularly from study start until at least 1 week after the last dose. Dyspepsia was monitored after esomeprazole withdrawal.

DETAILED DESCRIPTION:
Non-clinical studies have shown that PPI-induced hypergastrinaemia leads to rebound gastric hyperacidity after PPI withdrawal. A gastrin/CCK2 receptor antagonist inhibits that response. Studies in healthy subjects and patients also suggest that PPI withdrawal leads to rebound hyperacidity, but the evidence is controversial. However, there is better evidence from studies in healthy subjects that PPI withdrawal can lead to dyspepsia.

The principal aims of this study were: to assess the effect of different dose regimens of netazepide on the increases in circulating gastrin and CgA induced by esomeprazole in healthy subjects; and to choose a dose regimen for future studies of esomeprazole withdrawal in patients. The secondary aims were: to assess if omeprazole withdrawal leads to dyspepsia, and if so whether it can be prevented by netazepide; and to assess the likelihood of an interaction between esomeprazole and netazepide. Gastrin and CgA are biomarkers of acid suppression and increased ECL-cell activity, respectively.

This was a randomised, double-blind, placebo-controlled, parallel-group, pilot study, in which six groups of eight healthy subjects took esomeprazole 40 mg daily for 28 days, and netazepide 1, 5 or 25 mg, or placebo, daily during the last 14 days of esomeprazole dosing, or the 14 days immediately following esomeprazole withdrawal (25 mg only). Gastrin and CgA were measured before the start of dosing until at least one week after completion of dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men, post-menopausal women or pre-menopausal women, using one of the following methods of contraception: abstinence; condom and spermicide; intra-uterine device; or hysterectomy or tubal ligation
2. Age 18-75 years
3. A body mass index (Quetelet index) in the range 18.0-30.9 Body Mass Index = weight (kg)/height (m2)
4. Negative test for H. pylori
5. No history of dyspepsia symptoms
6. No history of peptic ulcer or oesophagitis
7. No history of treatment with a histamine H2 antagonist, proton pump inhibitor or antacid
8. Normal serum gastrin (no greater than 5% above the upper limit of the HMR laboratory reference range for gastrin)
9. Non-smokers or social smokers (defined as 10 or fewer cigarettes per week)
10. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial
11. Willingness to give written consent to participate after reading the Information and Consent Form, and after having the opportunity to discuss the trial with the investigator or delegate.

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Clinically relevant abnormal history, physical findings, ECG (> 450 msec), or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the subject.
3. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the subject's participation in the trial or make it unnecessarily hazardous.
4. Severe adverse reaction to any drug
5. Use, during the 14 days before the baseline visit, of a prescription medicine, especially one that inhibits or induces CYP3A4/5, CYP2C8 or CYP2C9, a hormone contraceptive and hormone replacement therapy.
6. Use, during the 14 days before the baseline visit, of herbal products, such as St John's wort.
7. Use of an over-the-counter medicine during the 7 days before the baseline visit, with the exception of paracetamol (up to 4 g daily).
8. Participation in another trial of a new chemical entity or a prescription medicine, or loss of more than 400 mL blood, within the previous 3 months.
9. Presence or history of drug or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Plasma chromogranin A (CgA) concentrations | 8 weeks
  We separated serum or plasma from blood, and stored samples at -20°C until assay by ELISA (serum gastrin: Immulite 2000, DPC. CV = 6.9%; plasma CgA: DAKO. CV = 7.2%) and validated HPLC/MS method (plasma netazepide: lower limit of quantification 0.5 ng/mL) (Redrup et al 2002).
Serum gastrin concentrations | 8 weeks
  We separated serum or plasma from blood, and stored samples at -20°C until assay by ELISA (serum gastrin: Immulite 2000, DPC. CV = 6.9%; plasma CgA: DAKO. CV = 7.2%) and validated HPLC/MS method (plasma netazepide: lower limit of quantification 0.5 ng/mL) (Redrup et al 2002).

SECONDARY OUTCOMES:
Dyspepsia scores | 8 weeks
  The dyspepsia questionnaire uses 4- or 5-point Likert scales to measure frequency and severity of 15 upper gastrointestinal symptoms, and the bother they cause (Talley et al 2001).
Antacid usage | 8 weeks
  Participants reported antacid usage.
Safety assessed by Vital signs, ECG variables, physical examinations, laboratory variables | 5 weeks
Tolerability assessed by Adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, Principal Investigator — Hammersmith Medicines Research

IPD SHARING:
Plan to Share IPD: No